CLINICAL TRIAL: NCT00808106
Title: Clinical, Cellular, and Molecular Investigations Into Oculocutaneous Albinism
Brief Title: Clinical, Cellular, and Molecular Investigation Into Oculocutaneous Albinism
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090035; 09-HG-0035
Record Dates: First submitted 2008-12-12; First posted 2008-12-15 (Estimated); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Oculocutaneous Albinism
Keywords: Oculocutaneous Albinism
MeSH Terms: conditions — Albinism, Oculocutaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Albinism: Patients with albinism

SUMMARY:
Oculocutaneous albinism (OCA) is a term used to describe inherited forms of hypopigmentation associated with 1) variable levels of cutaneous hypopigmentation, ocular hypopigmentation, and visual deficits, and 2) involvement of both of the major developmental types of pigmented cells, i.e., melanocytes and retinal pigment epithelium. OCA that affects only usually-pigmented tissues is termed isolated OCA. There are currently seven albinism types (OCA-1 to OCA-7). With the exception of OCA-5, eash is associated with a specific gene and is inherited in an autosomal recessive manner OCA-5 is a proposed type of albinism associated with the chromosomal location 4q24. OCA-1 results from defects in the enzyme tyrosinase, which catalyzes the rate-limiting step in melanin synthesis. The precise functions of the remaining genes are not yet fully understood, but several may be associated with the regulation of pH in the subcellular organelle where melanin in manufactured-the melanosome. The majority of persons with OCA have two pathogenic mutations identified in a known OCA-causing gene, but a substantial minority to not. Ocular albinism (OA) is an X-linked disorder caused by mutations in the GPR143 gene. It affects the eye in a manner similar to OCA, but has minimal or no skin manifestations.

In this protocol, we have four major goals:

1. To clinically and comprehensively characterize OCA types 1 - 7, and OA, with respect to the degree of hypopigmentation, genetic mutations, extent of ocular involvement, and longitudinal variation.
2. To use study participants cultured melanocytes to study pigment biology, variability in pigment formation related to genotype, and response to proposed treatments. Some of this work will be performed collaboratively.
3. To recruit study participants with hypopigmentation not due to known albinismcausing genes.
4. To evaluate methods of quantifying eye pigmentation, skin pigmentation and other clinical parameters that may be usable as outcome measures in future treatment studies.

To achieve those goals, we will perform clinical evaluations of persons with OCA and OA at the NIH Clinical Center; obtain cultured cells, plasma, serum and urine for future studies; and, perform mutation analysis on known OCA and/or OA genes and search for other genes responsible for albinism. Routine admissions will last 3 - 4 days and occur every 2 - 3 years.

DETAILED DESCRIPTION:
Oculocutaneous albinism (OCA) is a term used to describe inherited forms of hypopigmentation associated with 1) variable levels of cutaneous hypopigmentation, ocular hypopigmentation, and visual deficits, and 2) involvement of both of the major developmental types of pigmented cells, i.e., melanocytes and retinal pigment epithelium. OCA that affects

only usually-pigmented tissues is termed isolated OCA. There are currently seven albinism

types (OCA-1 to OCA-7). With the exception of OCA-5, eash is associated with a specific

gene and is inherited in an autosomal recessive manner (see Table 1). OCA-5 is a proposed

type of albinism associated with the chromosomal location 4q24. OCA-1 results from defects

in the enzyme tyrosinase, which catalyzes the rate-limiting step in melanin synthesis. The

precise functions of the remaining genes are not yet fully understood, but several may be

associated with the regulation of pH in the subcellular organelle where melanin in

manufactured the melanosome. The majority of persons with OCA have two pathogenic

mutations identified in a known OCA-causing gene, but a substantial minority to not. Ocular

albinism (OA) is an X-linked disorder caused by mutations in the GPR143 gene. It affects the

eye in a manner similar to OCA, but has minimal or no skin manifestations.

In this protocol, we have four major goals:

1. To clinically and comprehensively characterize OCA types 1 7, and OA, with respect

   to the degree of hypopigmentation, genetic mutations, extent of ocular involvement,

   and longitudinal variation.
2. To use study participants cultured melanocytes to study pigment biology, variability

   in pigment formation related to genotype, and response to proposed treatments. Some

   of this work will be performed collaboratively
3. To recruit study participants with hypopigmentation not due to known albinismcausing

   genes.
4. To evaluate methods of quantifying eye pigmentation, skin pigmentation and other

clinical parameters that may be usable as outcome measures in future treatment studies.

To achieve those goals, we will perform clinical evaluations of persons with OCA and OA at

the NIH Clinical Center; obtain cultured cells, plasma, serum and urine for future studies; and,

perform mutation analysis on known OCA and/or OA genes and search for other genes

responsible for albinism. Routine admissions will last 3 - 4 days and occur every 2 - 3 years.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients will be screened by requesting copies of the following materials at the time they contact the program:

1. An indication of ethnic background by the potential participant, which may be unknown .
2. Photographs of the potential participant that give an indication of skin complexion/pigmentation and undyed hair color (if available).
3. Ophthalmology or other visual specialist records documenting visual exam characteristics, potentially including iris transillumination, visual evoked potential and or characteristic eye findings (if available).
4. Genetic testing results (if available).

EXCLUSION CRITERIA:

Exclusion from the study will be made based on one or more of the following criteria:

1. Significant evidence that the potential participant has either OCA1A or OCA2 with a typical presentation, AND has an ethnic background that is wellrepresented in the current study (proportion in study exceeding the proportion in the United States population).

   The rationale for this exclusion is that: 1) from a biologicaland clinicalresearch perspective, we have an adequate number of OCA1A/

   OCA2 cases in the current study population; and 2) that, despite this, persons with ethnicities that are underrepresented in the study may inform our understanding of populationlevel molecular patterns in OCA1A/ OCA2 and cultural implications of albinism.
2. Persons who are under 1 year of age. This exclusion occurs because there is no urgency for a very early evaluation. Also, the Clinical Center staff and resources are more suited for the care of older children.
3. Persons who are too sick to travel safely to the NIH Clinical Center.
4. A judgment by the principal investigator that clinical resources are not available to enroll additional patients at any given time.
5. Persons who are currently incarcerated.
6. Adults who are incompetent to consent to the protocol.
7. Persons who have been diagnosed with a known nonoculocutaneous disorder of hypopigmentation such as HemanskyPudlak Syndrome, ChediakHigashi Syndrome, or Griscelli Syndrome.
8. Persons who have been diagnosed with a known disorder of focal hypopigmentation such as Waardenburg syndrome.

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with albinism
Sampling Method: Non-Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2008-12-11 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
A | Ongiong
  Collect data to refine existing knowledge about the range, course and severity of the visual, cutaneous, auditory and other potentialmanifestations of the various forms of OCA and of OA
B | Ongoing
  Conduct laboratory studies on patients cultured melanocytes and other biologic specimens to further understand the cell biology ofpigment formation relative to genetic mutation
C | Ongoing
  Pursue the discovery of novel molecular defects in patients who have albinism caused by mutations in pigmentation-related genes that have not yet been proven to be associated with human pigmentation disorders
D | Ongoing
  Search for and evaluate methods of quantifying eye pigmentation, skin pigmentation and other clinical parameters that may be usable as outcome measures in future treatment studies

CONTACTS AND LOCATIONS:
Overall Officials: David R Adams, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Goding CR. Melanocytes: the new Black. Int J Biochem Cell Biol. 2007;39(2):275-9. doi: 10.1016/j.biocel.2006.10.003. Epub 2006 Oct 7. PMID 17095283
- [Background] King RA, Pietsch J, Fryer JP, Savage S, Brott MJ, Russell-Eggitt I, Summers CG, Oetting WS. Tyrosinase gene mutations in oculocutaneous albinism 1 (OCA1): definition of the phenotype. Hum Genet. 2003 Nov;113(6):502-13. doi: 10.1007/s00439-003-0998-1. Epub 2003 Sep 10. PMID 13680365
- [Background] Creel D, O'Donnell FE Jr, Witkop CJ Jr. Visual system anomalies in human ocular albinos. Science. 1978 Sep 8;201(4359):931-3. doi: 10.1126/science.684419.
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2009-HG-0035.html